CLINICAL TRIAL: NCT05710250
Title: The Effects of Mindfulness Meditation on Brain Metabolism in the Limbic Regions Studied by Magnetic Resonance Spectroscopy; Correlations With the Memory Performance and Episodic Metamemetory of Students.
Acronym: MEMOREM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DR220244-MEMOREM; 2022-A02454-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness based stress reduction (MBSR) program (Experimental): 15 students will follow a 6-week MBSR program with 2h30 sessions per week in group and daily exercises lasting 30-40 minutes per day.
  Interventions: Behavioral: 6-week MBSR program
- Muscular relaxation program (Active Comparator): 15 students will follow a 6-week muscular relaxation program with 2h30 group sessions per week in group and daily exercises lasting 30-40 minutes per day.
  Interventions: Behavioral: 6-week muscular relaxation program

INTERVENTIONS:
Behavioral: 6-week MBSR program — Participants will follow a 6-week program of mindfulness meditation. MBSR teaches mindfulness meditation and mindful yoga exercises to develop non-judgmental awareness of moment-to-moment experience. The intervention duration is 6 weeks, with weekly two and half hours sessions. It will be delivered according to the fundamental concepts and specific techniques provided in the MBSR manualized protocol by Kabat-Zinn. The program also includes 30-min daily homework exercises.
  MBSR teaches four main mindfulness practices: (1) body scan, a process of moving attention through the body; (2) mindful movement, consisting of gentle yoga stretches to develop awareness of body in movement; (3) sitting meditation; and (4) walking meditation. Inquiry and didactic teaching is also a part of MBSR and allows for some detailed exploration of participants' experiences.
  Arms: Mindfulness based stress reduction (MBSR) program
Behavioral: 6-week muscular relaxation program — Control group : This group will follow a 6-week program of progressive muscle relaxation training in order to learn achieving a deep relaxation of the body through voluntary tensing and relaxing muscles. It proceeds by the individual sequentially tensing and then releasing specific groups of muscles throughout the body, and noticing how tension feels relative to relaxation.
  The accomplishment of physical relaxation promotes mental calmness in a parallel manner. This program is based on the work of Bernstein and Borkovec and Jacobson, and will be structured in 6-week group with weekly two and half hours sessions and out-of-session assignments for at-home practice (30-min daily).
  Arms: Muscular relaxation program

SUMMARY:
Stress reduction methods based on mindfulness meditation have been experiencing significant growth in various fields of society over the past twenty years. In the case of students, scientific work has shown that mindfulness training has a positive effect on their mental health and possibly on their academic performance through improved attention and memory. The effect of metamemory ("knowing what you know and what you don't know"), which plays an important part in students memorization and academic success, has not yet been explored.

Changes in brain structure have been noted by MRI in some regions after several weeks of mindfulness training, but very few studies have yet looked at changes in brain metabolism that can be observed by the spectrocopy technique.

The investigators will conduct a prospective randomized study with overall 30 female speech therapists student that will be enrolled and assigned randomly to two groups, in a 1:1 ratio : one groupe that will benefit from mindfulness training and the other group that will benefit from another method of stress reduction based on muscular relaxation.

The programs will extend over 6 weeks with session of 2h30 per week in groups having personnal daily exercices (30-40' per day). During the 3 weeks leading up to and the 2 weeks following the program, students will take tests exploring memory and metamemory, complete mental health questionnaires, and have a magnetic resonance imaging with spectroscopic analysis.

DETAILED DESCRIPTION:
The main objective of this study is to investigate the effects of a mindfulness based stress reduction (MBSR) program on the metabolism of regions involved in memorization (several limbic regions : hippocampus, amygdala, anterior and posterior cingulate)

The study also aims to :

1. Study the effects of MBSR program on memory and metamemory.
2. Study correlations between MBSR program effects on metamemory and scores on mental health scales (anxiety, depression, perceived stress, burnout)
3. Study the correlations between MBSR program effects on memory and metamemory with those on attentional capacities, working memory, executive functions and emotion regulation
4. Investigate the relationship between brain metabolites variations and the effect of the MBSR program on episodic memory and metamemory capacities, attention and emotions
5. Investigate the relationship between metabolite concentrations variations and variations in volume and thickness of the cortex.

ELIGIBILITY:
Inclusion Criteria:

Female

* Right-handed
* ≥ 18 years old
* Affiliated to a social security scheme
* Written consent signed by the participan

Exclusion Criteria:

* Inability to complete the entire study programme
* Previous participation in an MBSR or MBCT programme
* Current neurological pathology
* Current psychiatric pathology, score ≥ 3 on the PHQ-4 self-questionnaire
* Previous or ongoing psychological or psychiatric treatment
* Previous or current psychotropic treatment
* Usual contraindications to brain MRI (including claustrophobia, ocular metallic foreign body, pacemaker, neurostimulator, cochlear implants (or non-removable electronic medical equipment), old generation heart valves, vascular clips previously implanted on a cranial aneurysm).
* Pregnancy
* During the exclusion period of a clinical research study
* Under legal protection or deprived of liberty.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Glumatate concentrations (mM) at 8 Weeks | baseline and 8 weeks
  Glumatate concentrations (mM) are measured by magnetic resonance spectrocopy in left hippocampal formation

SECONDARY OUTCOMES:
Change in left hippocampal formation volumes (mm3) measured on MRI 3D T1w sequence | baseline and 8 weeks
Change in right amygdala volumes (mm3) measured on MRI 3D T1w sequence | baseline and 8 weeks
Change in posterior cingulate volumes (mm3) measured on MRI 3D T1w sequence | baseline and 8 weeks
Chang in overall brain volume measured on MRI 3D T1w sequence | baseline and 8 weeks
Change in score the Feeling of knowing task (FOK task) | baseline and 8 weks
  FOK task for episodic memory performance includes 4 distincts steps : (1) a learning phase of a 60 pairs of words, (2) a cued recall phase (number of correct recalls /60 ; number of incorrect recalls /60), (3) feeling of knowing phase, (4) recognition phase (number of correct recognition /60 ; number of incorrect recognition /60)
Change in score of the Trail Making Test (TMT) | baseline and 8 weeks
  TMT consists of two parts. In the first part (A), the subject must connect with a pen in the correct order 25 numbers from 1 to 25, which are distributed randomly.
  In the second part (B), the subject must connect with a pencil in the correct order an alternation of 13 numbers from 1 to 13 and 12 letters from A to L, which are also distributed randomly. The time in seconds to complete each part is measured.
Change in score of Stroop test | baseline and 8 weeks
  The test includes 3 phases. In each one, participant have to give maximum of correct answer.
  Score ranges from 0 to 100 for each phase
Change in score of N-Back test | Baseline and at 8 weeks
  Number of correct answer (yes or no). Total score /23
Change in score of attentional network test (ANT) | baseline and 8 weeks
  Test (ANT) is a computerized testing measure that analyses the three components of attention network : alerting, orienting, executive control.
  Each of these three attention components is measured in time.
Change in score of the number memory task | baseline and 8 weeks
  Number memory score in direct order, ranges from 0 to 16. Number memory score in indirect order, ranges from 0 to 16
Change in score of the Hospital Anxiety and Depression Scale (HADS) | baseline and 8 weeks
  Anxio-depressive symptomatology based on the HADS score. The questionnaire is divided in two subscales, one for anxiety and one for depression. Each subscore ranges from 0 to 21. Scores greater than or equal to 11 on either scale indicate anxious or depressive symptomatology.
Change in score of the Perceived Stress Scale (PSS) | baseline and 8 weeks
  Anxio-depressive symptomatology based on the PSS score. The total score ranges from 0 to 40. Higher scores reflect greater stress level.
Change in score of the Columbia Suicide Severity Rating Scale (C-SSRS) | baseline and 8 weeks
  Evaluation of suicidality through the C-SSRS. The suicidal ideation severity subscale ranges from 1 to 5 (with higher number indicating more severe ideation). The intensity of ideation subscale includes 5 questions each one ranging from 1 to 5 (with higher number indicating more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
Change in score of the World Health Organization Quality of Life (WHOQOL) | baseline and 8 weeks
  Quality of life based on the WHOQOL score. The total score ranges from 0 to 100. Higher scores reflect better health.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Philippe COTTIER, Principal Investigator — University hospital of Tours